CLINICAL TRIAL: NCT05880615
Title: Opioid Reduced Anesthesia With Parasternal CATheters on Postoperative Delirium After Cardiac Surgery
Acronym: ORACAT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN452022/CHUSTE
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Cardiac Disease
Keywords: Cardiac surgery; postoperative delirium; regional anesthesia; enhanced recovery after surgery
MeSH Terms: conditions — Heart Diseases; Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- opioid reduced anesthesia with parasternal catheters inserted before sternotomy: Patients with opioid reduced anesthesia with parasternal catheters inserted before sternotomy will be included.
  Interventions: Other: collection of datas
- Opioid Anesthesia (OA): Patients with Opioid Anesthesia (OA) will be included.
  Interventions: Other: collection of datas

INTERVENTIONS:
Other: collection of datas — collection of datas:
  * Post-operative occurrence (within the first 48 hours after extubation) of post-operative delirium via the CAM-ICU (Confusion Assessment Method for the Intensive Care Unit) scale result
  * Post-operative hypoxemia defined as a PaO2/FiO2 ratio < 300 in the first 48 hours after extubation
  * reflex ileus defined as the absence of gas and/or matter in the first 48 hours after extubation,
  * total morphine consumption in the first 48 hours after surgery
  * pain at 24 hours and 48 hours after surgery
  * post-operative nausea and vomiting, major complications (neurological, respiratory, cardiac, infectious)
  * mortality 30 days after surgery

SUMMARY:
PostOperative Delirium (POD) is the most common neuropsychiatric complication following cardiac surgery and may be related to morphine consumption. PostOperative Delirium (POD) prolongs hospital and intensive care unit (ICU) length of stay (LOS) and increases morbidity and mortality. No study has been conducted to demonstrate the effect of regional anesthesia using catheters inserted before sternotomy.

DETAILED DESCRIPTION:
This study investigate the effect of an enhanced recovery protocol using regional anesthesia on PostOperative Delirium (POD) onset.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Admitte for scheduled cardiac surgery with sternotomy under cardiopulmonary bypass (CPB) for coronary artery bypass grafting (CABG), surgical correction of valve disease (aortic, mitral or tricuspid) or combined surgery (coronary artery bypass grafting (CABG) and valve replacement).

Exclusion Criteria:

* Age over 85,
* emergency surgery or heart transplant,
* body mass index (BMI) more than 40 kg.m-2
* reoperation
* Renal insufficiency with glomerular filtration rate (GFR) less than 30 mL.min-1
* left ventricular ejection fraction less than 30%
* respiratory insufficiency with arterial pressure of oxygen less than 60 mmHg
* hepatic insufficiency with prothrombin rate less than 30% or cirrhosis
* chronic hyperglycemia not controlled
* pregnancy
* cognitive impairment chronic use of opioids or drug addiction
* epilepsy
* guardianship
* allergy to locals anesthesics or any drugs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Scheduled Cardiac Surgery for Coronary Artery Bypass Grafting or Valvular Sternotomy in Patients Aged 18 to 85 Years will be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Number of Postoperative delirium (POD) assessed using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) in the first 48 hours after surgery | Hours: 48
  assessed using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Delirium is diagnosed when criteria 1 and 2 are positive, as well as criteria 3 or 4.

SECONDARY OUTCOMES:
Number of hypoxemia postoperative in the first 48 hours after extubation | Hours: 48
  Data collected in medical record: PaO2/FiO2 < 300
Number of Ileus postoperative in the first 48 hours after extubation | Hours: 48
  Data collected in medical record:absence of gas and/or material
Total morphine consumption within 48h after extubation | Hours: 48
  Data collected in medical record
Pain at 24 hours and 48 hours postoperative | Hours: 24, 48
  Data collected in medical record
postoperative nausea and vomiting | Hours: 48
  Data collected in medical record.
major complications (neurological, respiratory, cardiac, infectious) | Hours: 48
  Data collected in medical record.
mortality at 30 days after surgery | Day: 30
  Data collected in medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie GRAND, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No